CLINICAL TRIAL: NCT07237438
Title: Total Intravenous Anesthesia Versus Balanced Anesthesia on Loss of Muscle Mass After Colorectal Cancer Surgery
Brief Title: TIVA Versus Balanced Anesthesia on Muscle Mass in CRC Surgery
Acronym: TIVABAL-CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: Regional Institute of Oncology, Iasi, Romania (Unknown)
Responsible Party: Principal Investigator, Ianis Siriopol, Lecturer, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 358/11.08.2025
Record Dates: First submitted 2025-09-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (CRC); Sarcopenia
Keywords: colorectal cancer; sarcopenia; ultrasound; bioimpedance
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total intravenous anaesthesia (Active Comparator)
  Interventions: Procedure: total intravenous anaesthesia
- sevoflurane anaesthesia (Active Comparator)
  Interventions: Procedure: sevoflurane anaesthesia

INTERVENTIONS:
Procedure: total intravenous anaesthesia — evaluate the impact of the type of anaesthesia (total intravenous anaesthesia (TIVA)/sevoflurane anaesthesia) for colorectal surgery on the muscle function and mass
  Arms: total intravenous anaesthesia
Procedure: sevoflurane anaesthesia — evaluate the impact of the type of anaesthesia (total intravenous anaesthesia (TIVA)/sevoflurane anaesthesia) for colorectal surgery on the muscle function and mass
  Arms: sevoflurane anaesthesia

SUMMARY:
This study is aimed at clarifying changes in body composition during the perioperative period and identifying risk factors for skeletal muscle mass loss in patients with colorectal cancer. The investigators will asess the impact of the type of anaesthesia (total intravenous anaesthesia/sevoflurane anaesthesia) for colorectal surgery on the muscle function and mass, which will be evaluated using ultrasound, dynamometry and bioimpedance.

ELIGIBILITY:
Inclusion Criteria:

• adult patients diagnosed with colorectal cancer and scheduled for open colorectal surgery at the Regional Institute of Oncology, Iaşi, Romania

Exclusion Criteria:

* lack the capacity to consent
* extremity amputation
* paraplegia
* diseases affecting the muscles (such as stroke, lower-limb immobilization from a plaster, neurodegenerative diseases, peripheral neuropathy or muscle dystrophy)
* terminal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic assessment of muscle mass | From enrollment to 5 days after surgery
  Ultrasonographic muscle assessment is standardised in the assessment of muscle according to the SARCUS (Sarcopenia through UltraSound) working group recommendations. Rectus femoris muscle will be evaluated at 50% distance between the anterior superior iliac spine and the superior pole of the patella, in a lying position with knees in 10°, for muscle thickness and muscle cross-sectional area (CSA). Three measurements will be taken for each data point, and the average value will be used for further analysis. The biceps brachii muscle will be evaluated at 50% distance acromioclavicular joint and the elbow crease, in a supine position. Muscle thickness can be easily defined as the maximal vertical distance between the superficial and deep fasciae.
Muscle function assessment | From enrollment to 5 days after surgery
  Measuring grip strength is simple and inexpensive. Grip strength will be determined bilaterally. Each measurement will be performed three times on the left and right extremities with 20 seconds intervals between the measurements. The maximum measured value in kilograms will be used for analysis.
Bioimpedance assessment of lean and fat tissue mass | From enrollment to 5 days after surgery
  The bioimpedance measurements will be performed by a trained operator according to the manufacturer's recommendations. The Body Composition Monitor provides a quantitative measure of lean tissue and fat tissue mass. In contrast to earlier bioimpedance methodologies, the bioimpedance spectroscopy expresses body composition as a three-compartment model, providing overhydration, lean tissue index (LTI), and fat tissue index (FTI), whereby LTI and FTI are the respective tissue masses normalized to height squared.

SECONDARY OUTCOMES:
Hospital length of stay | From enrollment to the patient discharge, up to 52 weeks
Mortality | 28 and 90-day mortality after surgery

OTHER OUTCOMES:
Correlation | From enrollment to 5 days after surgery
  Correlation between muscle strength and muscle mass using dynamometry and echography and bioimpedance at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Oncology, Iaşi, Romania, Iași, Romania

IPD SHARING:
Plan to Share IPD: Undecided